CLINICAL TRIAL: NCT01041079
Title: Laparoscopic Revision Gastric Bypass Surgery for Chronic Marginal Ulcers: a 10 Year Experience
Brief Title: Chronic Marginal Ulcers After Gastric Bypass
Acronym: ChronicMU
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Kelvin D Higa, MD; FACS; FASMBS; Professor of Surgery UCSF, UCSF Fresno / ALSA Medical Group, Inc. Minimally Invasive Surgery Program
Other Study IDs: CMC IRB No. 2008078; U1111-1112-9755 (Other: World Health Organization, Universal Trial Number)
Record Dates: First submitted 2009-12-25; First posted 2009-12-31 (Estimated); Last update posted 2010-01-01 (Estimated); Status verified 2009-12

CONDITIONS: Marginal Ulcer; Chronic Ulcer Disease; Persistent Ulcer Disease; Recurrent Ulcer Disease; Late Morbidity After Gastric Bypass
Keywords: ulcer disease; marginal ulcer; morbidity of gastric bypass; late morbidity of gastric bypass; chronic abdominal pain; GI hemorrhage; Perforation; Penetration; Obstruction
MeSH Terms: conditions — Peptic Ulcer; Gastrointestinal Hemorrhage; Bites and Stings

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chronic marginal ulcer after RYGB: Patients with intractable or chronic marginal ulcer disease after gastric bypass complaining of abdominal pain, GI bleeding, obstruction, perforation and penetration. Sometimes with other associated diagnosis such as narcotic and tobacco dependence, protein-calorie malnutrition, excessive weight loss, poor pouch emptying syndrome, weight regain, inadequate initial weight loss, severe dumping syndrome among others.

SUMMARY:
The purpose of this study is to determine the feasibility, safety, and efficacy of revision gastroplasty along with other adjunct procedures in the treatment of intractable / chronic marginal ulcers after Roux-en-Y gastric bypass. A secondary aim is the identification of good and poor outcome predictors after revisional strategies for intractable or chronic marginal ulcer.

DETAILED DESCRIPTION:
The epidemic of overweight and obesity in the United States of America along with its comorbidities continues to expand. Bariatric surgery has demonstrated to be the most effective and sustained method to control severe obesity and its comorbidities. For instance, type 2 diabetes mellitus was completely resolved in 76.8%, systemic arterial hypertension was resolved in 61.7%, dyslipidemia improved in 70% and obstructive sleep apnea-hypopnea syndrome was resolved in 85.7%. Furthermore, bariatric surgery significantly increases life expectancy (89%) and decreases overall mortality (30-40%), particularly deaths from diabetes, heart disease, and cancer. Lastly, preliminary evidence about downstream savings associated with bariatric surgery offset the initial costs in 2 to 4 years.

Since 1998, there has been a substantially progressive increase in bariatric surgery. In 2005, the ASMBS reported that 81% of bariatric procedures were approached laparoscopically and in 2007, 205,000 people had bariatric surgery in the United States from which approximately 80% of these were Gastric Bypass. Moreover, there is a mismatch between eligibility and receipt of bariatric surgery with just less than 1% of the eligible population being treated for morbid obesity through bariatric surgery. Along with the increasing number of elective primary weight loss procedures, up to 20% of post RYGB patients cannot sustain their weight loss beyond 2 to 3 years after the primary bariatric procedure. Thus, revisional surgery for poor weight loss and re-operations for technical or mechanical complications will rise in a parallel manner.

A common late complication after gastric bypass surgery is marginal ulceration, an ulcer at the margins of the gastrojejunostomy on the jejunal side. Its incidence after RYGB ranges from as low as 0.6 to as high as 16%. After 1,040 laparoscopic RYGB surgeries, the incidence rate, in our hands, is 1.4% and mainly related to NSAID´s use. In observational cohort studies, the presence of specific technical factors - staple-line dehiscence or gastro-gastric fistula, enlarged pouch, foreign material and local ischemia - and environmental factors - tobacco, NSAID´s, alcohol consumption, and H pylori infection among others - have been associated with marginal ulceration however the exact etiopathogenesis has not been completely elucidated.

Similar to peptic ulcer disease (PUD), most marginal ulcers respond to medical therapy, specifically sucralfate and acid-lowering medication. In contrast, when perforation, obstruction, penetration, bleeding and/or intractability presents, complex or complicated ulcer disease, warrants surgical intervention.

The intestinal mucosa is not typically exposed to gastric acid, which is neutralized by the alkaline biliopancreatic secretions. The jejunal mucosa has no natural barriers; when exposed to gastric acid, it ulcerates easily. Capella & Capella demonstrated that transecting the gastric segments significantly reduce staple-line dehiscence; this is the so-called divided gastric bypass. In the retrospective analysis of their consecutive series, the incidence for gastro-gastric fistula (GGF) formation after undivided gastric bypass (GBP) was 23%, after a partially divided GBP was 19%, after a completely divided GBP was 2% and after complete transection with interposition of the jejunal limb was 0% (p <0.001). MacLean et al confirmed that divided primary gastric bypass decreases GGF formation (29% vs. 3%). Also, patients who developed marginal ulcers had a lower pH as well as a greater time with a pH less than 2 correlating 100% with the presence of GGF; closure of the GGF increased the pH in the pouch with subsequent healing of the marginal ulcer.

An unusually large gastric pouch (such as horizontal pouches, retained fundus, long lesser curvature based pouches or enlarged after initially being sized adequately) contain more acid-producing parietal cells. Increased acid production in the pouch carries the risk of developing marginal ulcers. Acid secretion in the small pouch after RYGB is virtually absent. Smith et al measured basal and pentagastrin-stimulated gastric acid secretion from the pouch were significantly lower compared to age and sex-matched controls. Likewise, MacLean et al reported a significantly lower pH & greater time with pH <2 in the gastric pouches of marginal ulcers and/or GGF patients after RYGB compared to non-complicated RYGB controls. Thus, creating a esophagojejunostomy would solve the gastric acid factor for developing marginal ulcers however the high incidence of anastomotic failure and unknown weight loss results are prohibitive for this approach. Sapala et al created a micro-pouch or cardiojejunostomy to decrease at maximum the parietal cell mass with a low incidence of marginal ulcers (0.01% at 1 years of follow-up) as well as to limit the pouch dilation. By Histopathology with a semi-quantitative approach, Gustavsson et al reported less acid-producing parietal cells within smaller pouches. With his next study (n=12), Gustavsson et al, demonstrated a significantly higher time exposure to a pH<4 in patients with marginal ulcer after RYGB (4x3cm pouch) compared to controls (p< 0.01). Furthermore, after downsizing the pouch, repeated pH-metry showed the % of time with pH <4 declined from 100% prior to 6% after revisionary surgery.

The anastomotic techniques influence the incidence of marginal ulcers. Capella & Capella reported a consecutive series with significant decrement from 5.1% to 1.5% (p< 0.001) after switching from a stapled to a hand-sewn anastomosis. Likewise, after changing from an inner layer of absorbable suture and an outer layer of nonabsorbable material to a double-layer of absorbable suture the incidence rate improved from 1.6% to 0%. Dr Schauer´s group confirmed a significant improvement in the incidence rate of MU from a 2.6% with the use of nonabsorbable suture for the outer layer to 1.3% after the change to absorbable suture for both layers (p < 0.001).

Local ischemia, in the immediate postoperative period, is probably secondary to technical reasons. Fundamental aspects for decreasing tension and local ischemia at the gastrojejunostomy are dissection of the tissues around the pouch without devascularizing the lesser curvature and complete mobilization of a well-perfused Roux limb.

In epidemiological, clinical and experimental studies, NSAID´s have been identified as one of the three major risk factors for PUD. Wilson et al found NSAID´s consumption to significantly increase the risk for marginal ulcer following RYGB (adjusted OR 11.5, 95%CI 4.8-28).

In epidemiological, clinical and experimental studies, Tobacco is another major risk factor for PUD. Smoking carries an overall relative risk of 2.2 (95%CI, 2.0-2.3).

Helicobacter pylori (H pylori) infection carries an overall relative risk of 3.3 (95%CI, 2.6-4.4) for developing PUD. A synergistic relationship exists between H pylori infection and NSAID´s consumption for developing PUD with an overall risk of 3.5 (95%CI, 1.26-9.96) compared to either H pylori or NSAID´s negative individuals. In Papasavas et al study, preoperative H. pylori testing with prophylactic eradication did not decrease the incidence of MU or erosive pouch gastritis.

The pathophysiological mechanisms of damage to the gastric mucosa of ethanol and alcoholic beverages are poorly understood. There are no studies available about the effect of alcohol on marginal ulcer development after RYGB.

Cocaine use is responsible for approximately 143,000 Emergency Department visits annually; 19% of American, between 18 to 25 years old, have used cocaine: more than 1% of the Americans use cocaine at least once a week; and approximately 50% of all drug-related deaths were secondary to Cocaine. The temporal association between smoking cocaine (crack) and GI tract manifestations include ulceration, perforation, visceral infarction, and retroperitoneal fibrosis.

Re-operative strategies for addressing chronic marginal ulcers after gastric bypass have been scarcely described and mostly are reports of a case or small series of cases. The revisional strategies described are I) ulcer excision with revision of the gastrojejunostomy and gastric transection if needed, II) ulcer excision with pouch downsizing and redo of gastrojejunostomy, III) ulcer excision with resection of the ischemic Roux limb segment, and IV) ulcer excision and reversal. The possible adjuvant procedures includes I) proximal remnant gastrectomy (partial gastrectomy), and II) vagotomy.

In summary, there is scant information about late complications after gastric bypass especially after the widespread adoption of the laparoscopic approach and the modern anatomical construct of Roux-en-Y Gastric Bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Chronic/Intractable, either recurrent or persistent, marginal ulcers after Roux-en-Y gastric bypass surgery for clinically severe obesity

Exclusion Criteria:

* Chronic or Intractable marginal ulcer after other bariatric procedures
* Revision or re-operation by open approach
* missing records and/or unreachable patients with scant information for analysis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after Roux-en-Y gastric bypass for clinically severe obesity complicated with intractable or chronic marginal ulcer disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Morbidity and mortality | at discharge, 1 week, 3 weeks, 8 weeks, 3 months, 6 months, 1 year and annually thereafter for up to 4 years
Weight loss expressed as Body Mass Index and Percentage excess weight loss | at 6 months, 1 year and annually thereafter for up to 4 years
Remission or improvement of marginal ulcer-related symptoms | at 6 months, 1 year and annually thereafter for up to 4 years
Remission or improvement of comorbidities | at 6 months, 1 year and annually thereafter for up to 4 years

SECONDARY OUTCOMES:
Length of operative time which is defined as the time duration of operation measured in minutes from the first skin incision to the final closure of the skin incision | It is measured in minutes from the first skin incision to the final closure of the skin incision at the time of revisional surgery under study. It is a transoperative measure of outcome of the surgery under study
Length of Hospital Stay which is a measured of surgical recovery quantified and reported in days. It is a hospital pre-discharge traditional measure of outcome. | It is measured in days from the admission date to the discharge date for the hospitalization pertaining to revisional surgery under study.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Tercero, MD, Study Director — Research Associate, University of California San Francisco; Kelvin D Higa, MD, Principal Investigator — Professor of Surgery, University of California San Francisco
Locations (1):
- University of California San Francisco, Department of Surgery/Fresno Medical Education Program, Fresno, California, United States

REFERENCES:
- [Background] Higa KD, Boone KB, Ho T, Davies OG. Laparoscopic Roux-en-Y gastric bypass for morbid obesity: technique and preliminary results of our first 400 patients. Arch Surg. 2000 Sep;135(9):1029-33; discussion 1033-4. doi: 10.1001/archsurg.135.9.1029. PMID 10982506
- [Background] Hedley AA, Ogden CL, Johnson CL, Carroll MD, Curtin LR, Flegal KM. Prevalence of overweight and obesity among US children, adolescents, and adults, 1999-2002. JAMA. 2004 Jun 16;291(23):2847-50. doi: 10.1001/jama.291.23.2847. PMID 15199035
- [Background] McTigue KM, Harris R, Hemphill B, Lux L, Sutton S, Bunton AJ, Lohr KN. Screening and interventions for obesity in adults: summary of the evidence for the U.S. Preventive Services Task Force. Ann Intern Med. 2003 Dec 2;139(11):933-49. doi: 10.7326/0003-4819-139-11-200312020-00013. PMID 14644897
- [Background] Buchwald H, Avidor Y, Braunwald E, Jensen MD, Pories W, Fahrbach K, Schoelles K. Bariatric surgery: a systematic review and meta-analysis. JAMA. 2004 Oct 13;292(14):1724-37. doi: 10.1001/jama.292.14.1724. PMID 15479938
- [Background] Christou NV, Sampalis JS, Liberman M, Look D, Auger S, McLean AP, MacLean LD. Surgery decreases long-term mortality, morbidity, and health care use in morbidly obese patients. Ann Surg. 2004 Sep;240(3):416-23; discussion 423-4. doi: 10.1097/01.sla.0000137343.63376.19. PMID 15319713
- [Background] Adams TD, Gress RE, Smith SC, Halverson RC, Simper SC, Rosamond WD, Lamonte MJ, Stroup AM, Hunt SC. Long-term mortality after gastric bypass surgery. N Engl J Med. 2007 Aug 23;357(8):753-61. doi: 10.1056/NEJMoa066603. PMID 17715409
- [Background] Sjostrom L, Narbro K, Sjostrom CD, Karason K, Larsson B, Wedel H, Lystig T, Sullivan M, Bouchard C, Carlsson B, Bengtsson C, Dahlgren S, Gummesson A, Jacobson P, Karlsson J, Lindroos AK, Lonroth H, Naslund I, Olbers T, Stenlof K, Torgerson J, Agren G, Carlsson LM; Swedish Obese Subjects Study. Effects of bariatric surgery on mortality in Swedish obese subjects. N Engl J Med. 2007 Aug 23;357(8):741-52. doi: 10.1056/NEJMoa066254. PMID 17715408
- [Background] Cremieux PY, Buchwald H, Shikora SA, Ghosh A, Yang HE, Buessing M. A study on the economic impact of bariatric surgery. Am J Manag Care. 2008 Sep;14(9):589-96. PMID 18778174
- [Background] Santry HP, Gillen DL, Lauderdale DS. Trends in bariatric surgical procedures. JAMA. 2005 Oct 19;294(15):1909-17. doi: 10.1001/jama.294.15.1909. PMID 16234497
- [Background] Flum DR, Khan TV, Dellinger EP. Toward the rational and equitable use of bariatric surgery. JAMA. 2007 Sep 26;298(12):1442-4. doi: 10.1001/jama.298.12.1442. No abstract available. PMID 17895461
- [Background] Meguid MM, Glade MJ, Middleton FA. Weight regain after Roux-en-Y: a significant 20% complication related to PYY. Nutrition. 2008 Sep;24(9):832-42. doi: 10.1016/j.nut.2008.06.027. PMID 18725080
- [Background] Nguyen NT. Reoperations and revisions in bariatric surgery. Surg Endosc. 2007 Nov;21(11):1907-8. doi: 10.1007/s00464-007-9572-6. Epub 2007 Sep 8. No abstract available. PMID 17828427
- [Background] Sapala JA, Wood MH, Sapala MA, Flake TM Jr. Marginal ulcer after gastric bypass: a prospective 3-year study of 173 patients. Obes Surg. 1998 Oct;8(5):505-16. doi: 10.1381/096089298765554061. PMID 9819081
- [Background] Higa KD, Boone KB, Ho T. Complications of the laparoscopic Roux-en-Y gastric bypass: 1,040 patients--what have we learned? Obes Surg. 2000 Dec;10(6):509-13. doi: 10.1381/096089200321593706. PMID 11175957
- [Background] Sanyal AJ, Sugerman HJ, Kellum JM, Engle KM, Wolfe L. Stomal complications of gastric bypass: incidence and outcome of therapy. Am J Gastroenterol. 1992 Sep;87(9):1165-9. PMID 1519574
- [Background] Capella JF, Capella RF. Staple Disruption and Marginal Ulceration in Gastric Bypass Procedures for Weight Reduction. Obes Surg. 1996 Feb;6(1):44-49. doi: 10.1381/096089296765557259. PMID 10731249
- [Background] Capella JF, Capella RF. Gastro-gastric fistulas and marginal ulcers in gastric bypass procedures for weight reduction. Obes Surg. 1999 Feb;9(1):22-7; discussion 28. doi: 10.1381/096089299765553674. PMID 10065576
- [Background] Jordan JH, Hocking MP, Rout WR, Woodward ER. Marginal ulcer following gastric bypass for morbid obesity. Am Surg. 1991 May;57(5):286-8. PMID 2039124
- [Background] Sacks BC, Mattar SG, Qureshi FG, Eid GM, Collins JL, Barinas-Mitchell EJ, Schauer PR, Ramanathan RC. Incidence of marginal ulcers and the use of absorbable anastomotic sutures in laparoscopic Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2006 Jan-Feb;2(1):11-6. doi: 10.1016/j.soard.2005.10.013. PMID 16925306
- [Background] Lublin M, McCoy M, Waldrep DJ. Perforating marginal ulcers after laparoscopic gastric bypass. Surg Endosc. 2006 Jan;20(1):51-4. doi: 10.1007/s00464-005-0325-0. Epub 2005 Dec 7. PMID 16333541
- [Background] St Jean MR, Dunkle-Blatter SE, Petrick AT. Laparoscopic management of perforated marginal ulcer after laparoscopic Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2006 Nov-Dec;2(6):668. doi: 10.1016/j.soard.2006.09.011. No abstract available. PMID 17138240
- [Background] Chin EH, Hazzan D, Sarpel U, Herron DM. Multimedia article. Laparoscopic repair of a perforated marginal ulcer 2 years after gastric bypass. Surg Endosc. 2007 Nov;21(11):2110. doi: 10.1007/s00464-007-9486-3. Epub 2007 Aug 18. PMID 17704879
- [Background] Abstracts of the 2008 Scientific Session of the Society of American Gastrointestinal and Endoscopic Surgeons (SAGES), Philadelphia, Pennsylvania, USA, 9-12 April 2008. Surg Endosc. 2008 Apr;22 Suppl 1:144-301. doi: 10.1007/s00464-008-9821-3. No abstract available. PMID 18330642
- [Background] Nguyen NT, Hinojosa MW, Gray J, Fayad C. Reoperation for marginal ulceration. Surg Endosc. 2007 Nov;21(11):1919-21. doi: 10.1007/s00464-007-9538-8. Epub 2007 Aug 19. No abstract available. PMID 17705072
- [Background] Patel RA, Brolin RE, Gandhi A. Revisional operations for marginal ulcer after Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2009 May-Jun;5(3):317-22. doi: 10.1016/j.soard.2008.10.011. Epub 2008 Nov 6. PMID 19136312
- [Background] Madan AK, DeArmond G, Ternovits CA, Beech DJ, Tichansky DS. Laparoscopic revision of the gastrojejunostomy for recurrent bleeding ulcers after past open revision gastric bypass. Obes Surg. 2006 Dec;16(12):1662-8. doi: 10.1381/096089206779319400. PMID 17217644
- [Background] Huang JQ, Sridhar S, Hunt RH. Role of Helicobacter pylori infection and non-steroidal anti-inflammatory drugs in peptic-ulcer disease: a meta-analysis. Lancet. 2002 Jan 5;359(9300):14-22. doi: 10.1016/S0140-6736(02)07273-2. PMID 11809181
- [Background] Ramaswamy A, Lin E, Ramshaw BJ, Smith CD. Early effects of Helicobacter pylori infection in patients undergoing bariatric surgery. Arch Surg. 2004 Oct;139(10):1094-6. doi: 10.1001/archsurg.139.10.1094. PMID 15492150
- [Background] Rasmussen JJ, Fuller W, Ali MR. Marginal ulceration after laparoscopic gastric bypass: an analysis of predisposing factors in 260 patients. Surg Endosc. 2007 Jul;21(7):1090-4. doi: 10.1007/s00464-007-9285-x. Epub 2007 May 19. PMID 17514403
- [Background] Stenstrom B, Loseth K, Bevanger L, Sturegard E, Wadstrom T, Chen D. Gastric bypass surgery does not increase susceptibility to Helicobacter pylori infection in the stomach of rat or mouse. Inflammopharmacology. 2005;13(1-3):229-34. doi: 10.1163/156856005774423791. PMID 16259742
- [Background] Yang CS, Lee WJ, Wang HH, Huang SP, Lin JT, Wu MS. The influence of Helicobacter pylori infection on the development of gastric ulcer in symptomatic patients after bariatric surgery. Obes Surg. 2006 Jun;16(6):735-9. doi: 10.1381/096089206777346754. PMID 16756734
- [Background] Papasavas PK, Gagne DJ, Donnelly PE, Salgado J, Urbandt JE, Burton KK, Caushaj PF. Prevalence of Helicobacter pylori infection and value of preoperative testing and treatment in patients undergoing laparoscopic Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2008 May-Jun;4(3):383-8. doi: 10.1016/j.soard.2007.08.014. Epub 2007 Nov 5. PMID 17974495
- [Background] Teyssen S, Singer MV. Alcohol-related diseases of the oesophagus and stomach. Best Pract Res Clin Gastroenterol. 2003 Aug;17(4):557-73. doi: 10.1016/s1521-6918(03)00049-0. PMID 12828955
- [Background] Bode C, Bode JC. Effect of alcohol consumption on the gut. Best Pract Res Clin Gastroenterol. 2003 Aug;17(4):575-92. doi: 10.1016/s1521-6918(03)00034-9. PMID 12828956
- [Background] Glauser J, Queen JR. An overview of non-cardiac cocaine toxicity. J Emerg Med. 2007 Feb;32(2):181-6. doi: 10.1016/j.jemermed.2006.05.044. Epub 2007 Jan 22. PMID 17307630
- [Background] Lee HS, LaMaute HR, Pizzi WF, Picard DL, Luks FI. Acute gastroduodenal perforations associated with use of crack. Ann Surg. 1990 Jan;211(1):15-7. doi: 10.1097/00000658-199001000-00003. PMID 2403771
- [Background] Arrillaga A, Sosa JL, Najjar R. Laparoscopic patching of crack cocaine-induced perforated ulcers. Am Surg. 1996 Dec;62(12):1007-9. PMID 8955237
- [Background] Sharma R, Organ CH Jr, Hirvela ER, Henderson VJ. Clinical observation of the temporal association between crack cocaine and duodenal ulcer perforation. Am J Surg. 1997 Dec;174(6):629-32; discussion 632-3. doi: 10.1016/s0002-9610(97)00215-8. PMID 9409587
- [Background] Schuster KM, Feuer WJ, Barquist ES. Outcomes of cocaine-induced gastric perforations repaired with an omental patch. J Gastrointest Surg. 2007 Nov;11(11):1560-3. doi: 10.1007/s11605-007-0257-1. Epub 2007 Aug 15. PMID 17701263
- [Background] Mason EE. Warning patients about cocaine and aspirin. Obes Surg. 1998 Jun;8(3):312-3. doi: 10.1381/096089298765554539. No abstract available. PMID 9678199
- See also: "Click here for more information about the department sponsor´s web site" — http://www.fresno.ucsf.edu/surgery/